CLINICAL TRIAL: NCT07178535
Title: Feasibility of Two Types of Real-Time Visual Feedback in an Augmented Reality Environment to Reduce Spatial Gait Asymmetry in Adults Post-Stroke
Brief Title: Feasibility of Real-Time Visual Feedback in Augmented Reality to Reduce Gait Asymmetry Post-Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Anouk Lamontagne, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-50-2025-2284; 2025-2026 - BF7 - 363369 (Other Grant/Funding Number: FRQS)
Record Dates: First submitted 2025-09-03; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Post-stroke locomotor deficits; Spatial gait asymmetry; Real-time visual feedback; Augmented reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant (Experimental)
  Interventions: Device: Feasibility of Two Types of Real-Time Visual Feedback in an Augmented Reality

INTERVENTIONS:
Device: Feasibility of Two Types of Real-Time Visual Feedback in an Augmented Reality — Participants will walk in a corridor (45 m), equipped with "Xsens" inertial sensors recording their kinematics and an "HTC Vive Elite-XR" AR headset superimposing virtual feedback onto the real world. Three real-time feedback conditions (3 trials/condition) will be evaluated randomly: (1) an avatar reflecting the participant's movements; (2) visual bars indicating step lengths; (3) control condition without feedback. Participants take part in an evaluation/intervention session.

SUMMARY:
Unilateral motor deficits, such as paresis and tone disorders, are frequent consequences of stroke and lead to gait impairments. Among these, spatial asymmetry is characterized by differences in step length between the paretic and non-paretic limbs, resulting in balance problems and an increased risk of falls. Conventional rehabilitation has shown limited effectiveness in addressing this issue, highlighting the need for innovative approaches. Real-time feedback interventions, particularly through augmented reality (AR), may help improve gait asymmetry by providing a more natural and interactive learning environment.

This study aims to compare the effectiveness of two types of real-time visual feedback, an avatar-based system and visual bars, in improving gait symmetry and other locomotor parameters in individuals post-stroke. It will also assess the acceptability and usability of the intervention, participants' sense of presence, and the potential for cybersickness induced by these systems.

A repeated-measures design will be used to evaluate the immediate effectiveness of the two types of visual feedback on gait asymmetry and other locomotor parameters in adults in the subacute phase after stroke. Participants, aged 18 to 65 and presenting spatial asymmetry, will perform walking trials in an AR environment while being exposed to both feedback modalities in randomized order. Spatiotemporal and kinematic data will be collected using inertial sensors, while questionnaires will assess acceptability, usability, sense of presence, and cybersickness.

Participants will be evaluated in a 45-m long corridor (free of traffic) and will perform nine walking trials (three per condition) under three randomized conditions: (1) a lateral view avatar displayed on the paretic side, previously shown to provide optimal feedback on step length; (2) a visual bar feedback representing bilateral step lengths; and (3) a "control" condition with no additional feedback. Each walking trial, lasting 2.5 minutes, will consist of a pre-adaptation phase without feedback (30 s), followed by an adaptation phase with feedback (1 min), and a post-adaptation phase without feedback (1 min).

The investigators expect that avatar-based feedback will be more effective than visual bars in improving spatial symmetry. The investigators also anticipate that both feedback modalities will be well accepted and usable by participants without inducing cybersickness, but that the sense of presence will be higher with avatar-based feedback. This study will shed light on locomotor adjustment mechanisms and may lay the groundwork for future clinical trials. By offering a personalized, evidence-based approach, these results could help transform post-stroke rehabilitation through the integration of innovative tools to optimize functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be in the subacute phase, between 14 days and 6 months following a first supratentorial stroke
* able to walk with or without an assistive device for at least 2.5 minutes
* present spatial asymmetry (step length ratio, SLR > 1.08)

Exclusion Criteria:

* Abnormal or no-corrected visual acuity (EDTRS < 50/20)
* visual field deficits (Goldmann or computerized perimetry)
* cognitive impairment (Montreal Cognitive Assessment score < 22
* not being able to provide informed consent
* present other conditions besides stroke that limit walking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Step length ratio | For each condition the step length ratio will be assessed at each trial: before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  For the ratio calculation, the mean step length values from the left and right sides will be used, with the larger value placed in the numerator to ensure that all individual ratios are >1.0. A ratio of 1.0 will indicate perfect symmetry. We will compare the step length ratio (SLR)

SECONDARY OUTCOMES:
Walking speed | For each condition : before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  Comparison of walking speed (product of step length and cadence) in meter per second
Step width | For each condition : before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  Comparison of step width in meter
Gait cycle duration percentages | For each condition : before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  Gait cycle duration percentages (single support phase, corresponding to the contralateral swing phase, and double support phase) in percentage
Trunk and pelvis maximum range of motion | For each condition : before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  For the trunk and pelvis, we will measure the maximum range of motion in the sagittal and frontal planes in Degree
Hip and knee range of motion | For each condition : before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  For the hip and knee, we will measure in the sagittal plane the peak extension during stance, the peak flexion during swing, and the maximum range of motion. in Degree
Ankle range of motion | For each condition : before the pre-adaptation phase (T1: 0 s), after the pre-adaptation phase (T2: 0.5 min), after the adaptation phase (T3: 1.5 min), and after the post-adaptation phase (T4: 2.5 min).
  For the ankle, we will measure in the sagittal plane the peak dorsiflexion at initial contact and during swing, as well as the peak plantarflexion at the end of double support uring the gait cycle. In degree
Acceptability | Investigators will compare these parameters before et after the session.
  Participant's comments and observations collected using the Theoretical Framework of Acceptability (TFA) Questionnaire, which considers different dimensions such as affective attitude, perceived effectiveness, ethicality and opportunity cost. It comprises 8 items rated from 1 to 5. Minimum value is 8 and maximum value is 40. A higher score is associated with better outcomes.
Usability | Investigators will compare these parameters before and after the intervention.
  Participants' responses will be collected using the Single Ease Question (SEQ) questionnaire, which assesses task difficulty on a scale from 1 (very difficult) to 7 (very easy). The questionnaire consists of a single item, with higher scores indicating better usability.
Embodiment | Investigators will compare these parameters before et after the intervention.
  The Virtual Embodiment Questionnaire (VEQ) is a quantitative measure of the degree to which a person experiences a sense of embodiment in a virtual body within a virtual reality environment. The score is obtained by summing responses to the questionnaire items, which assess three key components of embodiment: body ownership (5 items), agency (5 items), and changes in body schema (6 items). For each item, participants indicate their level of agreement on a 7-point scale, where 1 corresponds to "strongly disagree" and 7 to "strongly agree." A higher score reflects a greater sense of virtual embodiment.
Sens of Presence | Investigators will compare these parameters before et after the session.
  The Holistic Presence Questionnaire (HPQ) is a quantitative measure of presence, assessing telepresence, internal and external plausibility, and perceived behavioral and cognitive affordances within a mediated environment in five items. For each item, participants indicate their level of agreement on a 7-point scale, where 1 corresponds to "strongly disagree" and 7 to "strongly agree." A higher score reflects a greater sense of presence in the virtual environment.
Cybersickness | Investigators will compare these parameters before et after the session
  The " Fast Motion Sickness Questionnaire " is a single-item verbal self-assessment scale ranging from 0 (no cybersickness) to 20 (severe cybersickness). A higher score indicates greater cybersickness

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish Rehabilitation Hospital - CISSS Laval, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided